CLINICAL TRIAL: NCT06225674
Title: A Retrospective, Observational, Post-market Clinical Investigation on the Outcome of Episealer Talus Post-operation for Treatment of Focal Osteochondral Defects
Brief Title: Clinical Investigation on the Outcome of Episealer Talus Post-operation for Treatment of Focal Osteochondral Defects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Episurf Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Epi_002
Record Dates: First submitted 2023-12-13; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Osteochondral Defect

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Episealer Talus implant — This is an observational study, no intervention will be done. The aim for the clinical investigation is to collect data from approximately 25 adult subjects who were treated for focal osteochondral defect with Episealer Talus implant in 6 clinics (Sweden and Germany) since January 2020.

SUMMARY:
This is a retrospective, observational, single-arm, multi-centre, post-market clinical investigation designed to verify clinical performance and safety of Episealer Talus post-operation for treatment of focal osteochondral defects on the talus bone in the ankle. This retrospective investigation aims to collect data from patients with focal osteochondral defects treated with Episealer Talus, to provide insight on the potential benefit of Episealer Talus in the treatment of focal osteochondral defects.

The aim for the clinical investigation is to collect data from approximately 25 adult subjects who were treated for focal osteochondral defect with Episealer Talus implant in 6 clinics (Sweden and Germany) since January 2020, when the devices were CE-marked. The data collected for each subject will include demographics and data generated in relation to the surgery itself and the post-surgery phases including e.g. focal defect grade and position, collected through medical record review. Each subject will also be asked to complete a set of QoL questionnaires (SEFAS, FAOS and VAS).

DETAILED DESCRIPTION:
This is a retrospective, observational, single-arm, multi-centre, post-market clinical investigation designed to verify clinical performance and safety of Episealer Talus post-operation for treatment of focal OCDs. The overall clinical investigation is based on the patient's reported outcome (PROs) from OCD patients previously treated with Episealer Talus implant after January 2020. In total approximately 25 adult subjects, male or female, from 6 clinics (Sweden and Germany) will be included in the investigation.

Subjects will be identified by the investigational site team through medical record review and/or site knowing the subjects from performing the implantation after January 2020. Following collection of the subject´s signed informed consent, subject demographics, health- and surgery-related data will be collected from the subjects' medical records. Therefore, only one visit is planned for each subject during the clinical investigation. The performance variables relate to quality of life, and all subjects will be asked to fill in three questionnaires (SEFAS, FAOS and VAS).

The overall duration of the investigation is estimated to be 4 months, including a 1 month recruitment period. Each subject is estimated to spend approximately 1-2 hour for completing the informed consent and completing the questionnaires. Subject´s participation in the clinical investigation will be terminated once the questionnaires have been completed and the site team considers all data collected for the subject.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Patients ≥ 18 years old at the time of index procedure
* Patients who previously received Episealer Talus implant after January 2020

Exclusion Criteria:

* "None"

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with Episealer Talus implant after January 2020. In total approximately 25 adult subjects, male or female, from 6 clinics (Sweden and Germany) will be included in the investigation.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2024-03-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of total SEFAS (self-reported foot and ankle score) outcome | 1 hour
  SEFAS data will be extracted from the patient´s reported outcome (PROs). Range 0-48, low score is better

SECONDARY OUTCOMES:
Assessment of total FAOS (Foot and Ankle Outcome Score) and subscale (pain, other symptoms, activities of daily living, sport and recreational function, | 30 minutes
  FAOS data will be extracted from the patient´s reported outcome (PROs). Range 0-100, low score is better
Assessment of total Visual Analogue Scale and subsections (rest, walking running, climb steps) | 10 minutes
  VAS data will be extracted from the patient´s reported outcome (PROs), Range 0-10, low score is better.
Surgery-related information | 10 minutes
  Retrospective data collection
Additional clinical performance parameters of Episealer Talus implant | 10 minutes
  Subject's and PI's treatment satisfaction (Self reported, scale 1-5 low score is better)

OTHER OUTCOMES:
The retrospective investigation design includes a non-systematic assessment of the spontaneous reporting of AEs, ADEs, SAEs, SADEs, and DDs. | 1 hour
  All safety variables, deriving from the non-systematic assessment, will be tabulated for the Safety Population: AE, ADE, SAE, SADE, and DD.

CONTACTS AND LOCATIONS:
Overall Officials: Jouko Kivioja, Principal Investigator — Aleris Hand @ Fot
Locations (6):
- Germany (4):
  - Robert-Koch-Krankenhaus Apolda, Apolda
  - OrthoCentrum Hamburg, Hamburg
  - St. Elisabeth-Krankenhaus, Salzgitter
  - St. Ansgar Sulingen-Bassum, Sulingen
- Sweden (2):
  - Aleris Hand @ Fot, Stockholm
  - FotCenter, Stockholm